CLINICAL TRIAL: NCT07118254
Title: A PHASE II PROSPECTIVE RANDOMIZED DOUBLE-MASKED CROSSOVER STUDY ASSESSING THE SAFETY & EFFICACY OF RHPRG4 (450 μG/ML RECOMBINANT HUMAN PROTEOGLYCAN 4) COMPARED TO VEHICLE FOR THE TREATMENT OF OCULAR GRAFT-VERSUS-HOST DISEASE (OGVHD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lubris Bio Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RHPRG4-oGVHD-002
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ocular Graft Versus Host Disease
Keywords: oGVHD; Dry Eye; Graft Versus Host Disease
MeSH Terms: conditions — Dry Eye Syndromes; Graft vs Host Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhPRG4 450ug/ml (Experimental): rhPRG4 450ug/ml
  Interventions: Drug: rhPRG4 450ug/ml
- Vehicle Control (Placebo Comparator): PBS Based Vehicle Control
  Interventions: Drug: Vehicle Control

INTERVENTIONS:
Drug: rhPRG4 450ug/ml — Treatment
  Arms: rhPRG4 450ug/ml
Drug: Vehicle Control — PBS Based Vehicle Control
  Arms: Vehicle Control

SUMMARY:
An 84-day, prospective, randomized (1:1) vehicle controlled, double-masked pre-market, crossover study. Subjects with moderate to severe oGVHD related Dry Eye Disease Each subject will receive both treatments in random sequence, each for 28 days, separated by a 14-day vehicle washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to comprehend and provide a signed and dated consent form.
2. Are 18-80 years of age at time of consent;
3. Have been diagnosed with oGVHD for at least 3 months prior to giving informed consent to participate in the trial;
4. Current use of artificial tears for the treatment of oGVHD related dry eye;
5. Have been stably using systemic medications for at least 14 days prior to Visit 1;
6. VAS Eye Dryness (100-point scale) score ≥ 40 mm;
7. Average VAS score for all symptoms of dry eye (dryness, foreign body sensation, burning/stinging, itching, pain, stick feeling, blurred vision and photophobia) ≥ 25 mm, none < 5 mm;
8. Have Oxford corneal fluorescein staining grade of ≥ 2 using the Oxford scale in the worst performing eye
9. Stated willingness to comply with all study procedures, attend all scheduled clinic visits, and continue participation for the duration of the study;
10. Ability to self-administer study medication and willingness to adhere to the medication regimen.

Exclusion Criteria:

Are currently or have a history of any ocular or systemic disorder or condition other than dry eye that based on investigator judgment will interfere with the interpretation of the study results. Examples of ocular or systemic disorders or conditions include active ocular infection, conjunctivochalasis, superior limbic keratoconjunctivitis, limbal stem cell deficiency, allergic conjunctivitis, giant papillary conjunctivitis, atopic keratoconjunctivitis, anterior basement membrane dystrophies, neurotrophic keratitis, corneal dystrophy, exposure keratitis, moderate to severe blepharitis, ocular trauma, progressive or degenerative corneal conditions, uveitis, and systemic infection; 2. History of any ocular surgery (including laser or refractive surgical procedures) or therapeutic medical devices in either eye within 30 days before study enrollment. Therapeutic medical devices include trigeminal stimulation, meibomian glad warming (excepting at home masks) or expression, intense pulsed light, low level light therapy, etc. Ocular surgeries include laser or refractive surgical procedures, insertion of punctal or punctal cauterization; Ocular surgery will not be allowed during study participation; 3. Initiation of new therapeutic modalities within 14 days of Visit 1; 4. Have a known hypersensitivity to one of the components of the study or procedural medications; 5. Have participated in another clinical study at the same time as the present study or within 30 days of the Visit 1; 6. Have a history of drug, medication or alcohol abuse or addiction; 7. Are females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) who meet any one of the following conditions:

1. are currently pregnant or,
2. have a positive result on the urine pregnancy test at the Screening/Baseline Visit or,
3. intend to become pregnant during the entire course of and 30 days after the study treatment periods, or,
4. are breast-feeding or,
5. not willing to use highly effective birth control measures, such as: hormonal contraceptives - oral, implanted, transdermal, or injected and/or mechanical barrier methods, during the entire course of and 30 days after the study treatment periods; 8. Per the discretion of the investigator or designee, history of a serious physical or mental disorder that prevents the subject from attending study visits, complying with study-related procedures, and/or prevents the subject's ability to make decisions on their own; 9. Any other surgical or medical condition or finding that in the opinion of the investigator would compromise the subject's safety or participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of rhPRG4 using the total corneal staining with fluorescein (Oxford Scale) compared to vehicle after 28 days of treatment | Baseline to day 28
  To assess the efficacy of rhPRG4 using the total corneal staining with fluorescein (Oxford Scale) compared to vehicle after 28 days of treatment
To assess the efficacy of rhPRG4 using the total VAS score (sum of dryness, foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision and photophobia, anchors: none & severe) compared to vehicle after 28 days of treatment | From baseline to day 28
  To assess the efficacy of rhPRG4 using the total VAS score (sum of dryness, foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision and photophobia, anchors: none & severe) compared to vehicle after 28 days of treatment

SECONDARY OUTCOMES:
To assess the efficacy of rhPRG4 using individual VAS scores for dryness, foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision and photophobia (anchors: none & severe) compared to vehicle after 28 days of treatment | From baseline to day 28
  To assess the efficacy of rhPRG4 using individual VAS scores for dryness, foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision and photophobia (anchors: none & severe) compared to vehicle after 28 days of treatment
To assess the efficacy of rhPRG4 using the SANDE score compared to vehicle after 28 days of treatment | From baseline to day 28
  To assess the efficacy of rhPRG4 using the SANDE score compared to vehicle after 28 days of treatment
To assess the efficacy of rhPRG4 using the maximum inter-eye tear osmolarity: max(OU) compared to vehicle after 28 days of treatment | From baseline to day 28
  To assess the efficacy of rhPRG4 using the maximum inter-eye tear osmolarity: max(OU) compared to vehicle after 28 days of treatment
To assess the safety of rhPRG4 by observation of the severity of treatment-emergent adverse events over the study duration | From baseline to day 28
  To assess the safety of rhPRG4 by observation of the severity of treatment-emergent adverse events over the study duration
To assess the safety of rhPRG4 by observation of the Best Corrected Distance Visual Acuity (BCVA) | From baseline to day 28
  To assess the safety of rhPRG4 by observation of the Best Corrected Distance Visual Acuity (BCVA)
To assess the safety of rhPRG4 by observation of signs evaluated by safety examination (ophthalmic examination plus slit lamp examination (SLE) of meibomian glands, eyelid Erythema, eyelid oedema, lashes, conjunctival erythema, lens, iris, anterior chamb | From baseline to day 28
  To assess the safety of rhPRG4 by observation of signs evaluated by safety examination (ophthalmic examination plus slit lamp examination (SLE) of meibomian glands, eyelid Erythema, eyelid oedema, lashes, conjunctival erythema, lens, iris, anterior chamber, hyperemia, corneal transparency & corneal neovascularization)
To assess the safety of rhPRG4 by observation of intraocular pressure (IOP) | From baseline to day 28
  To assess the safety of rhPRG4 by observation of intraocular pressure (IOP)

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Sydney Eye Hospital, Sydney, New South Wales
  - OTA, Brisbane, Queensland
  - Royal Melbourne Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided